CLINICAL TRIAL: NCT00454987
Title: Assessment of Long-term Antibody Persistence After a Booster Dose of GSK Biologicals' Hib & Meningococcal C Vaccine (Menitorix™) 811936 Given at 12-15 Months of Age to Subjects Primed With 3 Doses of Menitorix™ at 2, 3, 4 Months of Age
Brief Title: Study of Long-term Antibody Persistence After a Booster Dose of Menitorix Vaccine
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 109664; 109666 (Other: GSK); 109668 (Other: GSK); 2006-006460-32 (EudraCT Number)
Record Dates: First submitted 2007-03-30; First posted 2007-04-02 (Estimated); Results first posted 2015-12-16 (Estimated); Last update posted 2020-06-16 (Actual); Status verified 2020-06

CONDITIONS: Haemophilus Influenzae Type b; Neisseria Meningitidis; Neisseria Meningitidis-Haemophilus Influenzae Type b Vaccine
Keywords: antibody persistence; Meningococcal serogroup C vaccine; conjugate vaccine; Haemophilus influenzae type b vaccine
MeSH Terms: conditions — Haemophilus Infections

ARMS (3):
- Menitorix Group (Experimental): Previously primed in infancy with Menitorix™ and Infanrix-IPV™ and boosted with Menitorix™ (Priorix™ co-administered). All UK subjects received a booster dose of Infanrix-IPV™ at 40 to 43 months of age, intramuscularly in the deltoid region.
  Interventions: Biological: Infanrix IPV
- Meningitec Group (Active Comparator): Previously primed in infancy with Meningitec™ and Pediacel™ and boosted with Menitorix™ (Priorix™ co-administered). All UK subjects received a booster dose of Infanrix-IPV™ at 40 to 43 months of age, intramuscularly in the deltoid region.
  Interventions: Biological: Infanrix IPV
- Meningitec+Hiberix Group (Active Comparator): Previously primed (according to the routine UK immunisation schedule) with 3 doses of a Meningitec™ conjugate vaccine and a Hiberix™ containing vaccine before the age of 8 months without booster dose at 12 months of age (only for UK). All subjects received a booster dose of Infanrix-IPV™ and Menitorix™ at 40 to 43 months of age, intramuscularly in the deltoid region.
  This group was added only at year 2 in UK (Meningitec+Hiberix Group) to comply with UK Hib Catch-up vaccination programme.
  Interventions: Biological: Menitorix; Biological: Infanrix IPV

INTERVENTIONS:
Biological: Menitorix — Menitorix was only administered to subjects of the group Meningitic+Hiberix group at 40 to 43 months of age.
  Arms: Meningitec+Hiberix Group
Biological: Infanrix IPV — Infanrix IPV was administered according to the manufacturer's instructions to UK subjects at 40 to 43 months of age.

SUMMARY:
The purpose of this study is to evaluate the long-term antibody persistence at 12, 24 and 48 months after the administration of a booster dose of Menitorix™, given at 12-15 months of age. The children had previously received 3 doses of Menitorix™ and Infanrix IPV™ or Meningitec™ and Pediacel™ in infancy. In addition, the antibody persistence is to be investigated in children of 40-43 months of age who received a 3-dose primary vaccination of a MenC conjugate vaccine and a Hib containing vaccine in infancy without a booster dose of MenC conjugate and Hib vaccine in the second year of life.

This protocol posting deals with objectives & outcome measures of the extension phases at 12, 24 and 48 months after the booster phase. The links to objectives and outcome measures of the primary phase & booster phase at 12 to 15 months are provided below:

https://www.gsk-studyregister.com/study/2747 (Primary phase) https://www.gsk-studyregister.com/study/2755 (Booster phase)

DETAILED DESCRIPTION:
This multicentre & multicountry study is open and has 2 study groups at Visits 1 and 3 (HibMenC and LicMenC). An additional control group in the UK at the time of the second year follow-up for persistence (subjects aged 40-43 months primed with MenC conjugate and Hib vaccines in infancy with no subsequent booster dose, group NoBoost at Visit 2). These subjects will receive a Hib catch-up vaccine at 40-43 months of age. The subjects of groups HibMenC and LicMenC were randomized in the primary vaccination study 103974 and will not be further randomized. The subjects of group NoBoost will not be randomized. All subjects at the UK centre will receive Infanrix™-IPV at the second visit (i.e. 24 months after Menitorix booster or at 40-43 months of age). In addition, the subjects of group NoBoost will receive a Hib catch-up vaccine (Menitorix™) at the same visit.

Subjects of groups HibMenC and LicMenC will have 3 blood samples taken for immunogenicity analyses: at 12, 24 & 48 months after the booster vaccination. Subjects of group NoBoost will have 1 blood sample taken for immunogenicity analyses at 40-43 months of age. 75 new subjects will be enrolled in this study (group NoBoost).

ELIGIBILITY:
Inclusion Criteria:

Subjects of groups HibMenC and LicMenC at Visits 1, 2 and 3:

* Subjects who the investigator believes that their parents/guardians can and will comply with the requirements of the protocol.
* A male or female between and including 24 and 31 months of age at the time of Visit 1, between and including 40 and 43 months of age at Visit 2 and between and including 60 and 64 months at Visit 3.
* Written informed consent obtained from the parent or guardian of the subject.
* Healthy subjects as established by medical history and clinical examination before entering into the study.
* Having completed the booster vaccination study 104056.

Subjects of group NoBoost at Visit 2 (UK only):

* Subjects who the investigator believes that their parents/guardians can and will comply with the requirements of the protocol.
* A male or female between and including 40 and 43 months of age at Visit 2.
* Written informed consent obtained from the parent or guardian of the subject.
* Healthy subjects as established by medical history and clinical examination before entering into the study.
* Having received a 3-dose primary vaccination with a MenC conjugate vaccine and a Hib containing vaccine before the age of 8 months.

Exclusion Criteria:

* Previous administration of booster dose of Hib or meningococcal serogroup C except booster study vaccines during the study 104056.
* History of H. influenzae type b or meningococcal diseases.
* For UK subjects of groups HibMenC and LicMenC only: previous administration of a booster dose of a pertussis-containing vaccine except booster study vaccines during the study 104056.

Ages: 24 Months to 64 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 288 (Actual)
Dates: Start 2007-05-16 (Actual); Primary Completion 2007-10-12 (Actual); Study Completion 2007-10-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (9):
- Poland (8):
  - GSK Investigational Site, Bydgoszcz
  - GSK Investigational Site, Gdansk
  - GSK Investigational Site, Kielce
  - GSK Investigational Site, Krakow
  - GSK Investigational Site, Poznan
  - GSK Investigational Site, Siemianowice Śląskie
  - GSK Investigational Site, Trzebnica
  - GSK Investigational Site, Łęczna
- GSK Investigational Site, Oxford, Oxfordshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Khatami A, Snape MD, John T, Westcar S, Klinger C, Rollinson L, Boutriau D, Mesaros N, Wysocki J, Galaj A, Yu LM, Pollard AJ. Persistence of immunity following a booster dose of Haemophilus influenzae type B-Meningococcal serogroup C glycoconjugate vaccine: follow-up of a randomized controlled trial. Pediatr Infect Dis J. 2011 Mar;30(3):197-202. doi: 10.1097/INF.0b013e3181f728fd. PMID 20844459
- [Background] Khatami A, Snape MD, Wysocki J, John TM, Westcar S, Mesaros N, Peddiraju K, Boutriau D, Yu LM, Pollard AJ. Persistence of antibody response following a booster dose of Hib-MenC-TT glycoconjugate vaccine to five years: a follow-up study. Pediatr Infect Dis J. 2012 Oct;31(10):1069-73. doi: 10.1097/INF.0b013e318262528c. PMID 22673139
- [Background] Khatami A et al. Antibody concentrations against pertussis antigens at age 5 years following infant and pre-school immunisation: follow-on of a randomized controlled trial. Abstract presented at the 7th World Congress for World Society for Pediatric Infectious Diseases (WSPID). Melbourne, Australia, 16-19 November 2011.
- [Background] Khatami A et al. Persistence of antibody response following a booster dose of Hib-MenC-TT glycoconjugate vaccine: A phase IV open randomized controlled trial. Abstract presented at the 27th annual ESPID meeting, Brussels, Belgium, 9-13 June 2009.
- [Background] Snape MD et al. Persistence of antibody response following a booster dose of Hib-MenC-TT glycoconjugate vaccine to five years: a follow-on study. Abstract presented at the 7th World Congress for World Society for Pediatric Infectious Diseases (WSPID). Melbourne, Australia, 16-19 November 2011.
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Individual Participant Data Set: 109664 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 109664 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 109664 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 109664 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 109664 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study participant flow also includes data from the booster phase (NCT00258700), as SAEs were collected on all the subjects enrolled in the booster phase, which included subjects enrolled in the current NCT00454987 study.
Pre-assignment Details: Only subjects from booster phase who volunteered to participate in the long term follow up at year 1,2&4 were enrolled at the respective years,leading to higher enrolled subjects at year 2 (386) compared to year 1 (288)
Period: Booster Period (NCT00258700)
Arm/Group | Menitorix Group | Meningitec Group | Meningitec+Hiberix Group
Started | 359 | 117 | 0
Completed | 357 | 116 | 0
Not Completed | 2 | 1 | 0
Not completed — Adverse Event | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0
Period: Year 1 (NCT00454987)
Arm/Group | Menitorix Group | Meningitec Group | Meningitec+Hiberix Group
Started | 221 | 67 | 0
Completed | 221 | 67 | 0
Not Completed | 0 | 0 | 0
Period: Year 2 (NCT00454987)
Arm/Group | Menitorix Group | Meningitec Group | Meningitec+Hiberix Group
Started | 235 | 77 | 74
Completed | 235 | 77 | 74
Not Completed | 0 | 0 | 0
Period: Year 4 (NCT00454987)
Arm/Group | Menitorix Group | Meningitec Group | Meningitec+Hiberix Group
Started | 206 | 62 | 0
Completed | 206 | 62 | 0
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Menitorix Group | Meningitec Group | Meningitec+Hiberix Group | Total
Number analyzed (Participants) | 359 | 117 | 74 | 550
Age, Continuous [Mean (Standard Deviation); unit: Months] — Population: Age corresponds to year 1 data
  Months
    number analyzed (Participants) | 221 | 67 | 0 | 288
    (all) | 27.9 (0.97) | 27.7 (0.68) |  | 27.85 (0.91)
Age, Continuous [Mean (Standard Deviation); unit: Months] — Population: Baseline characteristic corresponds to year 2
  Months
    number analyzed (Participants) | 235 | 77 | 74 | 386
    (all) | 40.6 (0.76) | 40.6 (0.74) | 40.5 (0.71) | 40.5 (0.73)
Age, Continuous [Mean (Standard Deviation); unit: Months] — Population: Data presented for year 4
  Months
    number analyzed (Participants) | 206 | 62 | 0 | 268
    (all) | 61.1 (1.03) | 61.0 (1.25) |  | 61.0 (1.14)
Age, Continuous [Mean (Standard Deviation); unit: Months] — Population: Data presented corresponds to booster phase
  Months
    number analyzed (Participants) | 359 | 117 | 0 | 476
    (all) | 12.8 (0.75) | 12.8 (0.78) |  | 12.8 (0.76)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Data presented correspond to year 1
  Participants
    number analyzed (Participants) | 221 | 67 | 0 | 288
    Female | 114 | 33 |  | 147
    Male | 107 | 34 |  | 141
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Data presented for year 2
  Participants
    number analyzed (Participants) | 235 | 77 | 74 | 386
    Female | 117 | 37 | 28 | 182
    Male | 118 | 40 | 46 | 204
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Data presented for year 4
  Participants
    number analyzed (Participants) | 206 | 62 | 0 | 268
    Female | 102 | 31 |  | 133
    Male | 104 | 31 |  | 135
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Data presented corresponds to booster phase
  Participants
    number analyzed (Participants) | 359 | 117 | 0 | 476
    Female | 179 | 62 |  | 241
    Male | 180 | 55 |  | 235

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Serum Bactericidal Assay Using Baby Rabbit Complement (rSBA-MenC) Antibody Titers Equal to or Above 1:8
Description: The anti-meningococcal serogroup C activity was determined using a serum bactericidal test. The cut-off of the assay is a dilution of 1:8, resulting in 50% inhibition.
Time Frame: At Year 1
Population: The ATP cohort for persistence Year 1 included all evaluable subjects who received 3 doses of vaccines in study NCT00258700, who had available assay results for at least one tested antigen at Year 1.
Measure: Number; unit: Subjects
Arm/Group | Menitorix Group | Meningitec Group
Number analyzed (Participants) | 204 | 64
Subjects
  rSBA-MenC (Pre-Primary): number analyzed (Participants) | 204 | 60
  rSBA-MenC (Pre-Primary) | 12 | 3
  rSBA-MenC (Post-Primary): number analyzed (Participants) | 202 | 63
  rSBA-MenC (Post-Primary) | 200 | 63
  rSBA-MenC (Pre-Booster): number analyzed (Participants) | 202 | 62
  rSBA-MenC (Pre-Booster) | 163 | 39
  rSBA-MenC (Post-Booster): number analyzed (Participants) | 203 | 64
  rSBA-MenC (Post-Booster) | 201 | 61
  rSBA-MenC PIV (M12): number analyzed (Participants) | 200 | 59
  rSBA-MenC PIV (M12) | 178 | 41

2. Primary Outcome: Number of Subjects With rSBA-MenC Antibody Titers ≥ 1:128
Description: The anti-meningococcal serogroup C activity was determined using a serum bactericidal test. The cut-off of the assay is a dilution of 1:128, resulting in 50% inhibition.
Time Frame: At Year 1
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | Menitorix Group | Meningitec Group
Number analyzed (Participants) | 204 | 64
Subjects
  rSBA-MenC (Pre-Primary): number analyzed (Participants) | 204 | 60
  rSBA-MenC (Pre-Primary) | 3 | 0
  rSBA-MenC (Post-Primary): number analyzed (Participants) | 202 | 63
  rSBA-MenC (Post-Primary) | 189 | 63
  rSBA-MenC (Pre-Booster): number analyzed (Participants) | 202 | 62
  rSBA-MenC (Pre-Booster) | 94 | 19
  rSBA-MenC (Post-Booster): number analyzed (Participants) | 203 | 64
  rSBA-MenC (Post-Booster) | 199 | 56
  rSBA-MenC PIV (M12): number analyzed (Participants) | 200 | 59
  rSBA-MenC PIV (M12) | 109 | 17

3. Primary Outcome: rSBA-MenC Antibody Titers
Description: Antibody concentrations for the serogroup C serum bactericidal assay using baby rabbit complement were expressed as geometric mean titers (GMT) with 95% confidence intervals (CI). Titers bellow the cut-off of the test were given an arbitrary value of half the cut-off for the purpose of GMT calculation.
Time Frame: At Year 1
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titre
Arm/Group | Menitorix Group | Meningitec Group
Number analyzed (Participants) | 204 | 64
Titre
  rSBA-MenC (Pre-Primary): number analyzed (Participants) | 204 | 60
  rSBA-MenC (Pre-Primary) | 4.8 [4.3 to 5.3] | 4.3 [3.9 to 4.8]
  rSBA-MenC (Post-Primary): number analyzed (Participants) | 202 | 63
  rSBA-MenC (Post-Primary) | 624.7 [530.7 to 735.4] | 1000.0 [778.8 to 1284.2]
  rSBA-MenC (Pre-Booster): number analyzed (Participants) | 202 | 62
  rSBA-MenC (Pre-Booster) | 67.1 [52.8 to 85.3] | 32.4 [20.3 to 51.6]
  rSBA-MenC (Post-Booster): number analyzed (Participants) | 203 | 64
  rSBA-MenC (Post-Booster) | 2540.3 [2058.0 to 3135.5] | 517.4 [346.7 to 772.0]
  rSBA-MenC PIV (M12): number analyzed (Participants) | 200 | 59
  rSBA-MenC PIV (M12) | 123.0 [98.9 to 153.0] | 35.7 [23.4 to 54.5]

4. Primary Outcome: Number of Subjects With rSBA-MenC Antibody Titers ≥1:8
Description: as for outcome 1
Time Frame: At Year 2
Population: The ATP cohort for persistence Year 2 included for all evaluable subjects who received 3 doses of vaccines in study NCT00258700, with available results for at least one tested antigen at Year 2.
Measure: Number; unit: Subjects
Arm/Group | Menitorix Group | Meningitec Group
Number analyzed (Participants) | 228 | 76
Subjects
  rSBA-MenC (Pre-Primary): number analyzed (Participants) | 227 | 70
  rSBA-MenC (Pre-Primary) | 16 | 2
  rSBA-MenC (Post-Primary): number analyzed (Participants) | 224 | 73
  rSBA-MenC (Post-Primary) | 222 | 73
  rSBA-MenC (Pre-Booster): number analyzed (Participants) | 226 | 72
  rSBA-MenC (Pre-Booster) | 175 | 48
  rSBA-MenC (Post-Booster M1) | 227 | 73
  rSBA-MenC (Post-Booster M12): number analyzed (Participants) | 184 | 53
  rSBA-MenC (Post-Booster M12) | 164 | 37
  rSBA-MenC (Post-Booster M24): number analyzed (Participants) | 219 | 74
  rSBA-MenC (Post-Booster M24) | 147 | 30

5. Primary Outcome: Number of Subjects With rSBA-MenC Antibody Titers ≥ 1:8 for Meningitec+Hiberix Group
Description: as for outcome 1
Time Frame: At Year 2
Population: The ATP cohort for persistence Year 2 included all evaluable subjects who received 3 doses of Meningitec™ conjugate vaccine and a Hiberix™ vaccine before 8 months of age, with available results for at least one tested antigen at Year 2.
Measure: Number; unit: Subjects
Arm/Group | Meningitec+Hiberix Group
Number analyzed (Participants) | 68
Subjects | 30

6. Primary Outcome: Number of Subjects With rSBA-MenC Antibody Titers ≥ 1:128
Description: as for outcome 2
Time Frame: At Year 2
Population: as for outcome 4
Measure: Number; unit: Subjects
Arm/Group | Menitorix Group | Meningitec Group
Number analyzed (Participants) | 228 | 76
Subjects
  rSBA-MenC (Pre-Primary): number analyzed (Participants) | 227 | 70
  rSBA-MenC (Pre-Primary) | 5 | 0
  rSBA-MenC (Post-Primary): number analyzed (Participants) | 224 | 73
  rSBA-MenC (Post-Primary) | 208 | 73
  rSBA-MenC (Pre-Booster): number analyzed (Participants) | 226 | 72
  rSBA-MenC (Pre-Booster) | 96 | 22
  rSBA-MenC (Post-Booster M1) | 225 | 66
  rSBA-MenC (Post-Booster M12): number analyzed (Participants) | 184 | 53
  rSBA-MenC (Post-Booster M12) | 98 | 15
  rSBA-MenC (Post-Booster M24): number analyzed (Participants) | 219 | 74
  rSBA-MenC (Post-Booster M24) | 86 | 10

7. Primary Outcome: Number of Subjects With rSBA-MenC Antibody Titers ≥ 1:128 for Meningitec+Hiberix Group
Description: as for outcome 2
Time Frame: At Year 2
Population: The ATP cohort for persistence Year 2 included for all evaluable subjects who received 3 doses of a Meningitec™ conjugate vaccine and a Hiberix™ vaccine before 8 months of age, with available results for at least one tested antigen at Year 2.
Measure: Number; unit: Subjects
Arm/Group | Meningitec+Hiberix Group
Number analyzed (Participants) | 68
Subjects | 11

8. Primary Outcome: rSBA-MenC Antibody Titers
Description: Antibody concentrations for anti-serogroup C serum bactericidal assay using baby rabbit complement were expressed as geometric mean titers (GMT) with 95% confidence intervals (CI). Titers below the cut-off of the test were given an arbitrary value of half the cut-off for the purpose of GMT calculation.
Time Frame: At Year 2
Population: The ATP cohort for persistence Year 2 included all evaluable subjects who received 3 doses of vaccines in study NCT00258700, with available results for at least one tested antigen at Year 2.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Menitorix Group | Meningitec Group
Number analyzed (Participants) | 228 | 76
Titer
  rSBA-MenC (Pre-Primary): number analyzed (Participants) | 227 | 70
  rSBA-MenC (Pre-Primary) | 5.0 [4.4 to 5.6] | 4.2 [3.9 to 4.5]
  rSBA-MenC (Post-Primary): number analyzed (Participants) | 224 | 73
  rSBA-MenC (Post-Primary) | 592.3 [507.3 to 691.5] | 1075.6 [859.8 to 1345.5]
  rSBA-MenC (Pre-Booster): number analyzed (Participants) | 226 | 72
  rSBA-MenC (Pre-Booster) | 58.6 [46.4 to 73.9] | 35.0 [23.1 to 53.0]
  rSBA-MenC (Post-Booster M1) | 2320.8 [1926.2 to 2796.2] | 520.9 [367.9 to 737.6]
  rSBA-MenC (Post-Booster M12): number analyzed (Participants) | 184 | 53
  rSBA-MenC (Post-Booster M12) | 122.3 [97.5 to 153.4] | 35.9 [22.9 to 56.0]
  rSBA-MenC (Post-Booster M24): number analyzed (Participants) | 219 | 74
  rSBA-MenC (Post-Booster M24) | 48.0 [36.8 to 62.6] | 14.4 [9.7 to 21.6]

9. Primary Outcome: rSBA-MenC Antibody Titers for Meningitec+Hiberix Group
Description: Antibody concentrations for anti-serogroup C serum bactericidal assay using baby rabbit complement were expressed as geometric mean titers (GMT) with 95% confidence intervals (CI). Titers bellow the cut-off of the test were given an arbitrary value of half the cut-off for the purpose of GMT calculation.
Time Frame: At Year 2
Population: The ATP cohort for persistence Year 2 included all evaluable subjects who received 3 doses of a Meningitec™ conjugate vaccine and a Hiberix™ vaccine before 8 months of age, with available results for at least one tested antigen at Year 2.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Meningitec+Hiberix Group
Number analyzed (Participants) | 68
Titer | 15.9 [10.3 to 24.3]

10. Primary Outcome: Number of Subjects With rSBA-MenC Antibody Titers ≥ 1:8
Description: as for outcome 1
Time Frame: At Year 4
Population: The ATP cohort for persistence Year 4 included all evaluable subjects who received 3 doses of vaccines in study NCT00258700, who had assay results available for at least one tested antigen at Year 4.
Measure: Number; unit: Subjects
Arm/Group | Menitorix Group | Meningitec Group
Number analyzed (Participants) | 195 | 58
Subjects
  rSBA-MenC (Pre-Primary): number analyzed (Participants) | 194 | 53
  rSBA-MenC (Pre-Primary) | 10 | 2
  rSBA-MenC (Post-Primary): number analyzed (Participants) | 194 | 55
  rSBA-MenC (Post-Primary) | 192 | 55
  rSBA-MenC (Pre-Boost): number analyzed (Participants) | 195 | 55
  rSBA-MenC (Pre-Boost) | 156 | 34
  rSBA-MenC (Post-Boost M1) | 194 | 56
  rSBA-MenC (Post-Boost M12): number analyzed (Participants) | 166 | 45
  rSBA-MenC (Post-Boost M12) | 148 | 30
  rSBA-MenC (Post-Boost M24): number analyzed (Participants) | 187 | 56
  rSBA-MenC (Post-Boost M24) | 123 | 20
  rSBA-MenC (Post-Boost M48): number analyzed (Participants) | 194 | 58
  rSBA-MenC (Post-Boost M48) | 115 | 26

11. Primary Outcome: Number of Subjects With rSBA-MenC Antibody Titers ≥ 1:128
Description: as for outcome 2
Time Frame: At Year 4
Population: as for outcome 10
Measure: Number; unit: Subjects
Arm/Group | Menitorix Group | Meningitec Group
Number analyzed (Participants) | 195 | 58
Subjects
  rSBA-MenC (Pre-Primary): number analyzed (Participants) | 194 | 53
  rSBA-MenC (Pre-Primary) | 2 | 0
  rSBA-MenC (Post-Primary): number analyzed (Participants) | 194 | 55
  rSBA-MenC (Post-Primary) | 182 | 55
  rSBA-MenC (Pre-Boost): number analyzed (Participants) | 195 | 55
  rSBA-MenC (Pre-Boost) | 87 | 17
  rSBA-MenC (Post-Boost M1) | 193 | 50
  rSBA-MenC (Post-Boost M12): number analyzed (Participants) | 166 | 45
  rSBA-MenC (Post-Boost M12) | 88 | 11
  rSBA-MenC (Post-Boost M24): number analyzed (Participants) | 187 | 56
  rSBA-MenC (Post-Boost M24) | 78 | 6
  rSBA-MenC (Post-Boost M48): number analyzed (Participants) | 194 | 58
  rSBA-MenC (Post-Boost M48) | 58 | 5

12. Primary Outcome: rSBA-MenC Antibody Titers
Description: as for outcome 9
Time Frame: At Year 4
Population: as for outcome 10
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Menitorix Group | Meningitec Group
Number analyzed (Participants) | 195 | 58
Titer
  rSBA-MenC (Pre-Primary): number analyzed (Participants) | 194 | 53
  rSBA-MenC (Pre-Primary) | 4.7 [4.2 to 5.2] | 4.2 [3.9 to 4.6]
  rSBA-MenC (Post-Primary): number analyzed (Participants) | 194 | 55
  rSBA-MenC (Post-Primary) | 616.1 [521.3 to 728.2] | 983.9 [742.6 to 1303.7]
  rSBA-MenC (Pre-Boost): number analyzed (Participants) | 195 | 55
  rSBA-MenC (Pre-Boost) | 64.3 [50.3 to 82.4] | 30.8 [18.8 to 50.4]
  rSBA-MenC (Post-Boost M1) | 2537.0 [2071.9 to 3106.5] | 507.0 [338.3 to 759.8]
  rSBA-MenC (Post-Boost M12): number analyzed (Participants) | 166 | 45
  rSBA-MenC (Post-Boost M12) | 124.1 [97.5 to 158.0] | 30.6 [18.7 to 50.1]
  rSBA-MenC (Post-Boost M24): number analyzed (Participants) | 187 | 56
  rSBA-MenC (Post-Boost M24) | 47.9 [35.7 to 64.3] | 12.1 [7.7 to 18.8]
  rSBA-MenC (Post-Boost M48): number analyzed (Participants) | 194 | 58
  rSBA-MenC (Post-Boost M48) | 30.4 [22.9 to 40.4] | 11.3 [7.7 to 16.5]

13. Primary Outcome: Number of Subjects With Anti-polyribosylribitol Phosphate (Anti-PRP) Antibodies Equal to or Above 0.15 Micrograms Per Milliliter (µg/mL) and Equal to or Above 1 Micrograms Per Milliliter (µg/mL)
Description: The anti-polyribosylribitol phosphate was determined using an Enzyme-linked Immunosorbent Assay (ELISA).
Time Frame: At Year 1
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | Menitorix Group | Meningitec Group
Number analyzed (Participants) | 206 | 64
Subjects
  Anti-PRP ≥ 0.15 µg/mL (Pre-Primary): number analyzed (Participants) | 206 | 63
  Anti-PRP ≥ 0.15 µg/mL (Pre-Primary) | 84 | 25
  Anti-PRP ≥ 1.0 µg/mL (Pre-Primary): number analyzed (Participants) | 206 | 63
  Anti-PRP ≥ 1.0 µg/mL (Pre-Primary) | 204 | 58
  Anti-PRP ≥ 0.15 µg/mL (Post-Primary): number analyzed (Participants) | 204 | 63
  Anti-PRP ≥ 0.15 µg/mL (Post-Primary) | 199 | 45
  Anti-PRP ≥ 1.0 µg/mL (Post-Primary): number analyzed (Participants) | 204 | 63
  Anti-PRP ≥ 1.0 µg/mL (Post-Primary) | 203 | 63
  Anti-PRP ≥ 0.15 µg/mL (Pre-Boost): number analyzed (Participants) | 204 | 64
  Anti-PRP ≥ 0.15 µg/mL (Pre-Boost) | 198 | 63
  Anti-PRP ≥ 1.0 µg/mL (Pre-Boost): number analyzed (Participants) | 204 | 64
  Anti-PRP ≥ 1.0 µg/mL (Pre-Boost) | 20 | 11
  Anti-PRP ≥ 0.15 µg/mL (Post-Boost): number analyzed (Participants) | 203 | 63
  Anti-PRP ≥ 0.15 µg/mL (Post-Boost) | 198 | 43
  Anti-PRP ≥ 1.0 µg/mL (Post-Boost): number analyzed (Participants) | 203 | 63
  Anti-PRP ≥ 1.0 µg/mL (Post-Boost) | 120 | 19
  Anti-PRP ≥ 0.15 µg/mL PIV (M12): number analyzed (Participants) | 198 | 63
  Anti-PRP ≥ 0.15 µg/mL PIV (M12) | 203 | 63
  Anti-PRP ≥ 1.0 µg/mL PIV (M12): number analyzed (Participants) | 198 | 63
  Anti-PRP ≥ 1.0 µg/mL PIV (M12) | 188 | 52

14. Primary Outcome: Concentration of Anti-PRP Antibodies
Description: Antibody concentrations for anti-polyribosylribitol phosphate were expressed as geometric mean concentrations (GMC) with 95% confidence intervals (CI), given in µg/mL. Concentrations bellow the cut-off of the test were given an arbitrary value of half the cut-off for the purpose of GMC calculation.
Time Frame: At Year 1
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | Menitorix Group | Meningitec Group
Number analyzed (Participants) | 206 | 64
µg/mL
  Anti-PRP (Pre-Primary): number analyzed (Participants) | 206 | 63
  Anti-PRP (Pre-Primary) | 0.160 [0.137 to 0.186] | 0.178 [0.130 to 0.243]
  Anti-PRP (Post-Primary): number analyzed (Participants) | 204 | 63
  Anti-PRP (Post-Primary) | 12.413 [10.688 to 14.417] | 2.473 [1.557 to 3.928]
  Anti-PRP (Pre-Boost): number analyzed (Participants) | 204 | 64
  Anti-PRP (Pre-Boost) | 1.293 [1.095 to 1.528] | 0.441 [0.309 to 0.627]
  Anti-PRP (Post-Boost): number analyzed (Participants) | 203 | 63
  Anti-PRP (Post-Boost) | 88.667 [74.609 to 105.373] | 39.024 [30.588 to 49.786]
  Anti-PRP PIV (M12): number analyzed (Participants) | 198 | 63
  Anti-PRP PIV (M12) | 7.153 [6.029 to 8.486] | 3.162 [2.316 to 4.318]

15. Primary Outcome: Number of Subjects With Anti-PRP Antibodies ≥ 0.15 µg/mL and ≥ 1 µg/mL
Description: The anti-polyribosylribitol phosphate was determined using an Enzyme-linked Immunosorbent Assay (ELISA).
Time Frame: At Year 2
Population: as for outcome 8
Measure: Number; unit: Subjects
Arm/Group | Menitorix Group | Meningitec Group
Number analyzed (Participants) | 230 | 75
Subjects
  Anti-PRP ≥ 0.15 µg/mL (Pre-Primary): number analyzed (Participants) | 230 | 73
  Anti-PRP ≥ 0.15 µg/mL (Pre-Primary) | 93 | 30
  Anti-PRP ≥ 1.0 µg/mL (Pre-Primary): number analyzed (Participants) | 230 | 73
  Anti-PRP ≥ 1.0 µg/mL (Pre-Primary) | 18 | 9
  Anti-PRP ≥ 0.15 µg/mL (Post-Primary): number analyzed (Participants) | 227 | 73
  Anti-PRP ≥ 0.15 µg/mL (Post-Primary) | 227 | 66
  Anti-PRP ≥ 1.0 µg/mL (Post-Primary): number analyzed (Participants) | 227 | 73
  Anti-PRP ≥ 1.0 µg/mL (Post-Primary) | 222 | 52
  Anti-PRP ≥ 0.15 µg/mL (Pre-Boost): number analyzed (Participants) | 229 | 74
  Anti-PRP ≥ 0.15 µg/mL (Pre-Boost) | 222 | 53
  Anti-PRP ≥ 1.0 µg/mL (Pre-Boost): number analyzed (Participants) | 229 | 74
  Anti-PRP ≥ 1.0 µg/mL (Pre-Boost) | 134 | 21
  Anti-PRP ≥ 0.15 µg/mL (Post-Boost M1): number analyzed (Participants) | 228 | 75
  Anti-PRP ≥ 0.15 µg/mL (Post-Boost M1) | 228 | 75
  Anti-PRP ≥ 1.0 µg/mL (Post-Boost M1): number analyzed (Participants) | 228 | 75
  Anti-PRP ≥ 1.0 µg/mL (Post-Boost M1) | 228 | 75
  Anti-PRP ≥ 0.15 µg/mL (Post-Boost M12): number analyzed (Participants) | 182 | 57
  Anti-PRP ≥ 0.15 µg/mL (Post-Boost M12) | 182 | 57
  Anti-PRP ≥ 1.0 µg/mL (Post-Boost M12): number analyzed (Participants) | 182 | 57
  Anti-PRP ≥ 1.0 µg/mL (Post-Boost M12) | 172 | 48
  Anti-PRP ≥ 0.15 µg/mL (Post-Boost M24): number analyzed (Participants) | 228 | 75
  Anti-PRP ≥ 0.15 µg/mL (Post-Boost M24) | 227 | 74
  Anti-PRP ≥ 1.0 µg/mL (Post-Boost M24): number analyzed (Participants) | 228 | 75
  Anti-PRP ≥ 1.0 µg/mL (Post-Boost M24) | 203 | 56

16. Primary Outcome: Number of Subjects With Anti-PRP Antibodies ≥0.15 µg/mL and ≥1 µg/mL for Meningitec+Hiberix Group
Description: The anti-polyribosylribitol phosphate was determined using an Enzyme-linked Immunosorbent Assay (ELISA).
Time Frame: At Year 2
Population: as for outcome 5
Measure: Number; unit: Subjects
Arm/Group | Meningitec+Hiberix Group
Number analyzed (Participants) | 72
Subjects
  Anti-PRP ≥ 0.15 µg/mL (Aged 40-43 mths) | 62
  Anti-PRP ≥ 1.0 µg/mL (Aged 40-43 mths) | 28

17. Primary Outcome: Concentration of Anti-PRP Antibodies
Description: Antibody concentrations for anti-polyribosylribitol phosphate were expressed as geometric mean concentrations (GMC) with 95% confidence intervals (CI), given in µg/mL. Concentrations below the cut-off of the test were given an arbitrary value of half the cut-off for the purpose of GMC calculation.
Time Frame: At Year 2
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | Menitorix Group | Meningitec Group
Number analyzed (Participants) | 230 | 75
µg/mL
  Anti-PRP (Pre-Primary): number analyzed (Participants) | 230 | 73
  Anti-PRP (Pre-Primary) | 0.153 [0.134 to 0.176] | 0.163 [0.125 to 0.213]
  Anti-PRP (Post-Primary): number analyzed (Participants) | 227 | 73
  Anti-PRP (Post-Primary) | 12.794 [11.159 to 14.669] | 2.396 [1.580 to 3.635]
  Anti-PRP (Pre-Boost): number analyzed (Participants) | 229 | 74
  Anti-PRP (Pre-Boost) | 1.260 [1.080 to 1.469] | 0.425 [0.310 to 0.582]
  Anti-PRP (Post-Boost M1): number analyzed (Participants) | 228 | 75
  Anti-PRP (Post-Boost M1) | 91.981 [78.700 to 107.503] | 44.002 [34.546 to 56.048]
  Anti-PRP (Post-Boost M12): number analyzed (Participants) | 182 | 57
  Anti-PRP (Post-Boost M12) | 7.107 [5.931 to 8.516] | 3.456 [2.488 to 4.799]
  Anti-PRP (Post-Boost M24): number analyzed (Participants) | 228 | 75
  Anti-PRP (Post-Boost M24) | 4.790 [4.065 to 5.644] | 2.339 [1.798 to 3.042]

18. Primary Outcome: Concentration of Anti-PRP Antibodies for Meningitec+Hiberix Group
Description: as for outcome 17
Time Frame: At Year 2
Population: as for outcome 5
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | Meningitec+Hiberix Group
Number analyzed (Participants) | 72
µg/mL | 0.668 [0.467 to 0.956]

19. Primary Outcome: Number of Subjects With Anti-PRP Antibodies ≥ 0.15 µg/mL and ≥ 1 µg/mL
Description: The anti-polyribosylribitol phosphate was determined using an Enzyme-linked Immunosorbent Assay (ELISA).
Time Frame: At Year 4
Population: as for outcome 10
Measure: Number; unit: Subjects
Arm/Group | Menitorix Group | Meningitec Group
Number analyzed (Participants) | 197 | 58
Subjects
  Anti-PRP ≥ 0.15 µg/mL (Pre-Primary): number analyzed (Participants) | 197 | 56
  Anti-PRP ≥ 0.15 µg/mL (Pre-Primary) | 77 | 24
  Anti-PRP ≥ 1.0 µg/mL (Pre-Primary): number analyzed (Participants) | 197 | 56
  Anti-PRP ≥ 1.0 µg/mL (Pre-Primary) | 14 | 9
  Anti-PRP ≥ 0.15 µg/mL (Post-Primary): number analyzed (Participants) | 196 | 55
  Anti-PRP ≥ 0.15 µg/mL (Post-Primary) | 196 | 48
  Anti-PRP ≥ 1.0 µg/mL (Post-Primary): number analyzed (Participants) | 196 | 55
  Anti-PRP ≥ 1.0 µg/mL (Post-Primary) | 191 | 33
  Anti-PRP ≥ 0.15 µg/mL (Pre-Boost): number analyzed (Participants) | 197 | 57
  Anti-PRP ≥ 0.15 µg/mL (Pre-Boost) | 191 | 38
  Anti-PRP ≥ 1.0 µg/mL (Pre-Boost): number analyzed (Participants) | 197 | 57
  Anti-PRP ≥ 1.0 µg/mL (Pre-Boost) | 119 | 14
  Anti-PRP ≥ 0.15 µg/mL (Post-Boost M1): number analyzed (Participants) | 195 | 57
  Anti-PRP ≥ 0.15 µg/mL (Post-Boost M1) | 195 | 57
  Anti-PRP ≥ 1.0 µg/mL (Post-Boost M1): number analyzed (Participants) | 195 | 57
  Anti-PRP ≥ 1.0 µg/mL (Post-Boost M1) | 195 | 57
  Anti-PRP ≥ 0.15 µg/mL (Post-Boost M12): number analyzed (Participants) | 164 | 48
  Anti-PRP ≥ 0.15 µg/mL (Post-Boost M12) | 164 | 48
  Anti-PRP ≥ 1.0 µg/mL (Post-Boost M12): number analyzed (Participants) | 164 | 48
  Anti-PRP ≥ 1.0 µg/mL (Post-Boost M12) | 157 | 40
  Anti-PRP ≥ 0.15 µg/mL (Post-Boost M24): number analyzed (Participants) | 194 | 56
  Anti-PRP ≥ 0.15 µg/mL (Post-Boost M24) | 193 | 55
  Anti-PRP ≥ 1.0 µg/mL (Post-Boost M24): number analyzed (Participants) | 194 | 56
  Anti-PRP ≥ 1.0 µg/mL (Post-Boost M24) | 174 | 40
  Anti-PRP ≥ 0.15 µg/mL (Post-Boost M48) | 197 | 58
  Anti-PRP ≥ 1.0 µg/mL (Post-Boost M48) | 171 | 36

20. Primary Outcome: Concentration of Anti-PRP Antibodies
Description: as for outcome 17
Time Frame: At Year 4
Population: as for outcome 10
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | Menitorix Group | Meningitec Group
Number analyzed (Participants) | 197 | 58
µg/mL
  Anti-PRP (Pre-Primary): number analyzed (Participants) | 197 | 56
  Anti-PRP (Pre-Primary) | 0.149 [0.129 to 0.173] | 0.180 [0.130 to 0.250]
  Anti-PRP (Post-Primary): number analyzed (Participants) | 196 | 55
  Anti-PRP (Post-Primary) | 12.715 [10.945 to 14.771] | 1.776 [1.058 to 2.979]
  Anti-PRP (Pre-Boost): number analyzed (Participants) | 197 | 57
  Anti-PRP (Pre-Boost) | 1.276 [1.080 to 1.508] | 0.380 [0.263 to 0.550]
  Anti-PRP (Post-Boost M1): number analyzed (Participants) | 195 | 57
  Anti-PRP (Post-Boost M1) | 90.101 [76.087 to 106.697] | 39.105 [29.506 to 51.825]
  Anti-PRP (Post-Boost M12): number analyzed (Participants) | 164 | 48
  Anti-PRP (Post-Boost M12) | 7.455 [6.176 to 8.998] | 3.557 [2.450 to 5.165]
  Anti-PRP (Post-Boost M24): number analyzed (Participants) | 194 | 56
  Anti-PRP (Post-Boost M24) | 4.928 [4.135 to 5.873] | 2.083 [1.524 to 2.847]
  Anti-PRP (Post-Boost M48) | 3.824 [3.218 to 4.543] | 1.673 [1.215 to 2.305]

21. Primary Outcome: Number of Subjects With Anti-serogroup C Polysaccharide (Anti-PSC) Antibody Concentrations Equal to or Above 0.3 Micrograms Per Milliliter(µg/mL) and Equal to or Above 2 Micrograms Per Milliliter (µg/mL)
Description: The anti-polysaccharide C activity was determined using an Enzyme-linked Immunosorbent Assay (ELISA).
Time Frame: At Year 1
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | Menitorix Group | Meningitec Group
Number analyzed (Participants) | 206 | 64
Subjects
  Anti-PSC ≥ 0.3 µg/mL (Pre-Primary): number analyzed (Participants) | 206 | 63
  Anti-PSC ≥ 0.3 µg/mL (Pre-Primary) | 19 | 4
  Anti-PSC ≥ 2 µg/mL (Pre-Primary): number analyzed (Participants) | 206 | 63
  Anti-PSC ≥ 2 µg/mL (Pre-Primary) | 8 | 1
  Anti-PSC ≥ 0.3 µg/mL (Post-Primary): number analyzed (Participants) | 202 | 63
  Anti-PSC ≥ 0.3 µg/mL (Post-Primary) | 202 | 63
  Anti-PSC ≥ 2 µg/mL (Post-Primary): number analyzed (Participants) | 202 | 63
  Anti-PSC ≥ 2 µg/mL (Post-Primary) | 201 | 63
  Anti-PSC ≥ 0.3 µg/mL (Pre-Booster): number analyzed (Participants) | 201 | 64
  Anti-PSC ≥ 0.3 µg/mL (Pre-Booster) | 170 | 56
  Anti-PSC ≥ 2 µg/mL (Pre-Booster): number analyzed (Participants) | 201 | 64
  Anti-PSC ≥ 2 µg/mL (Pre-Booster) | 27 | 10
  Anti-PSC ≥ 0.3 µg/mL (Post-Booster): number analyzed (Participants) | 205 | 64
  Anti-PSC ≥ 0.3 µg/mL (Post-Booster) | 205 | 64
  Anti-PSC ≥ 2 µg/mL (Post-Booster): number analyzed (Participants) | 205 | 64
  Anti-PSC ≥ 2 µg/mL (Post-Booster) | 183 | 47
  Anti-PSC ≥ 0.3 µg/mL (PIV [M12]): number analyzed (Participants) | 193 | 59
  Anti-PSC ≥ 0.3 µg/mL (PIV [M12]) | 119 | 29
  Anti-PSC ≥ 2 µg/mL (PIV [M12]): number analyzed (Participants) | 193 | 59
  Anti-PSC ≥ 2 µg/mL (PIV [M12]) | 19 | 2

22. Primary Outcome: Concentration of Anti-PSC Antibodies
Description: Antibody concentrations for anti-polysaccharide C were expressed as geometric mean concentrations (GMC) with 95% confidence intervals (CI), given in µg/mL. Concentrations bellow the cut-off of the test were given an arbitrary value of half the cut-off for the purpose of GMC calculation.
Time Frame: At Year 1
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | Menitorix Group | Meningitec Group
Number analyzed (Participants) | 206 | 64
µg/mL
  Anti-PSC (Pre-Primary): number analyzed (Participants) | 206 | 63
  Anti-PSC (Pre-Primary) | 0.18 [0.17 to 0.20] | 0.17 [0.15 to 0.18]
  Anti-PSC (Post-Primary): number analyzed (Participants) | 202 | 63
  Anti-PSC (Post-Primary) | 9.52 [8.68 to 10.45] | 11.20 [9.42 to 13.33]
  Anti-PSC (Pre-Booster): number analyzed (Participants) | 201 | 64
  Anti-PSC (Pre-Booster) | 0.77 [0.67 to 0.88] | 0.84 [0.66 to 1.06]
  Anti-PSC (Post-Booster): number analyzed (Participants) | 205 | 64
  Anti-PSC (Post-Booster) | 7.36 [6.46 to 8.39] | 3.51 [2.84 to 4.32]
  Anti-PSC (PIV [M12]): number analyzed (Participants) | 193 | 59
  Anti-PSC (PIV [M12]) | 0.47 [0.40 to 0.55] | 0.32 [0.26 to 0.40]

23. Primary Outcome: Number of Subjects With Anti-PSC Antibody Concentrations ≥ 0.3 µg/mL and ≥ 2 µg/mL
Description: The anti-polysaccharide C activity was determined using an Enzyme-linked Immunosorbent Assay (ELISA).
Time Frame: At Year 2
Population: as for outcome 4
Measure: Number; unit: Subjects
Arm/Group | Menitorix Group | Meningitec Group
Number analyzed (Participants) | 230 | 76
Subjects
  Anti-PSC ≥ 0.3 µg/mL (Pre-Primary): number analyzed (Participants) | 229 | 73
  Anti-PSC ≥ 0.3 µg/mL (Pre-Primary) | 26 | 6
  Anti-PSC ≥ 2 µg/mL (Pre-Primary): number analyzed (Participants) | 229 | 73
  Anti-PSC ≥ 2 µg/mL (Pre-Primary) | 12 | 1
  Anti-PSC ≥ 0.3 µg/mL (Post-Primary): number analyzed (Participants) | 225 | 72
  Anti-PSC ≥ 0.3 µg/mL (Post-Primary) | 225 | 72
  Anti-PSC ≥ 2 µg/mL (Post-Primary): number analyzed (Participants) | 225 | 72
  Anti-PSC ≥ 2 µg/mL (Post-Primary) | 224 | 72
  Anti-PSC ≥ 0.3 µg/mL (Pre-Booster): number analyzed (Participants) | 226 | 74
  Anti-PSC ≥ 0.3 µg/mL (Pre-Booster) | 188 | 66
  Anti-PSC ≥ 2 µg/mL (Pre-Booster): number analyzed (Participants) | 226 | 74
  Anti-PSC ≥ 2 µg/mL (Pre-Booster) | 27 | 13
  Anti-PSC ≥ 0.3 µg/mL (Post-Booster [M1] | 230 | 76
  Anti-PSC ≥ 2 µg/mL (Post-Booster) [M1] | 210 | 59
  Anti-PSC ≥ 0.3µg/mL (Post-Booster [M12]: number analyzed (Participants) | 178 | 54
  Anti-PSC ≥ 0.3µg/mL (Post-Booster [M12] | 110 | 26
  Anti-PSC ≥ 2 µg/mL (Post-Booster [M12]): number analyzed (Participants) | 178 | 54
  Anti-PSC ≥ 2 µg/mL (Post-Booster [M12]) | 16 | 2
  Anti-PSC ≥0.3 µg/mL (Post-Booster [M24]: number analyzed (Participants) | 226 | 75
  Anti-PSC ≥0.3 µg/mL (Post-Booster [M24] | 76 | 17
  Anti-PSC ≥ 2 µg/mL (Post-Booster [M24]): number analyzed (Participants) | 226 | 75
  Anti-PSC ≥ 2 µg/mL (Post-Booster [M24]) | 5 | 0

24. Primary Outcome: Number of Subjects With Anti-PSC Antibody Concentrations ≥ 0.3 µg/mL and ≥ 2 µg/mL for Meningitec+Hiberix Group
Description: The anti-polysaccharide C activity was determined using an Enzyme-linked Immunosorbent Assay (ELISA).
Time Frame: At Year 2
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Meningitec+Hiberix Group
Number analyzed (Participants) | 72
Participants
  Anti-PSC ≥ 0.3 µg/mL (Aged 40-43 mths) | 4
  Anti-PSC ≥2 µg/mL (Aged 40-43 mths) | 0

25. Primary Outcome: Concentration of Anti-PSC Antibodies
Description: as for outcome 22
Time Frame: At Year 2
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | Menitorix Group | Meningitec Group
Number analyzed (Participants) | 230 | 76
µg/mL
  Anti-PSC (Pre-Primary): number analyzed (Participants) | 229 | 73
  Anti-PSC (Pre-Primary) | 0.20 [0.18 to 0.22] | 0.17 [0.15 to 0.18]
  Anti-PSC (Post-Primary): number analyzed (Participants) | 225 | 72
  Anti-PSC (Post-Primary) | 9.35 [8.56 to 10.22] | 12.29 [10.50 to 14.39]
  Anti-PSC (Pre-Booster): number analyzed (Participants) | 226 | 74
  Anti-PSC (Pre-Booster) | 0.74 [0.65 to 0.84] | 0.87 [0.69 to 1.10]
  Anti-PSC (Post-Booster [M1]) | 7.41 [6.59 to 8.33] | 3.91 [3.19 to 4.79]
  Anti-PSC (Post-Booster [M12]): number analyzed (Participants) | 178 | 54
  Anti-PSC (Post-Booster [M12]) | 0.47 [0.40 to 0.55] | 0.32 [0.25 to 0.40]
  Anti-PSC (Post-Booster [M24]): number analyzed (Participants) | 226 | 75
  Anti-PSC (Post-Booster [M24]) | 0.25 [0.23 to 0.28] | 0.21 [0.18 to 0.24]

26. Primary Outcome: Concentration of Anti-PSC Antibodies for Meningitec+Hiberix Group
Description: as for outcome 22
Time Frame: At Year 2
Population: as for outcome 5
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | Meningitec+Hiberix Group
Number analyzed (Participants) | 72
µg/mL | 0.16 [0.15 to 0.18]

27. Primary Outcome: Number of Subjects With Anti-PSC Antibody Concentrations ≥ 0.3 µg/mL and ≥ 2 µg/mL
Description: The anti-polysaccharide C activity was determined using an Enzyme-linked Immunosorbent Assay (ELISA).
Time Frame: At Year 4
Population: as for outcome 10
Measure: Number; unit: Subjects
Arm/Group | Menitorix Group | Meningitec Group
Number analyzed (Participants) | 197 | 58
Subjects
  Anti-PSC ≥ 0.3 µg/mL (Pre-Primary): number analyzed (Participants) | 197 | 56
  Anti-PSC ≥ 0.3 µg/mL (Pre-Primary) | 19 | 3
  Anti-PSC ≥ 2 µg/mL (Pre-Primary): number analyzed (Participants) | 197 | 56
  Anti-PSC ≥ 2 µg/mL (Pre-Primary) | 7 | 1
  Anti-PSC ≥ 0.3 µg/mL (Post-Primary): number analyzed (Participants) | 197 | 54
  Anti-PSC ≥ 0.3 µg/mL (Post-Primary) | 194 | 54
  Anti-PSC ≥ 2 µg/mL (Post-Primary): number analyzed (Participants) | 197 | 54
  Anti-PSC ≥ 2 µg/mL (Post-Primary) | 193 | 54
  Anti-PSC ≥ 0.3 µg/mL (Pre-Boost): number analyzed (Participants) | 197 | 57
  Anti-PSC ≥ 0.3 µg/mL (Pre-Boost) | 163 | 52
  Anti-PSC ≥ 2 µg/mL (Pre-Boost): number analyzed (Participants) | 194 | 57
  Anti-PSC ≥ 2 µg/mL (Pre-Boost) | 24 | 9
  Anti-PSC ≥ 0.3 µg/mL (Post-Boost [M1]) | 197 | 58
  Anti-PSC ≥ 2 µg/mL (Post-Boost [M1]) | 179 | 43
  Anti-PSC ≥ 0.3 µg/mL (Post-Boost [M12]): number analyzed (Participants) | 161 | 45
  Anti-PSC ≥ 0.3 µg/mL (Post-Boost [M12]) | 101 | 22
  Anti-PSC ≥ 2 µg/mL (Post-Boost [M12]): number analyzed (Participants) | 161 | 45
  Anti-PSC ≥ 2 µg/mL (Post-Boost [M12]) | 15 | 2
  Anti-PSC ≥ 0.3 µg/mL (Post-Boost [M24]): number analyzed (Participants) | 193 | 56
  Anti-PSC ≥ 0.3 µg/mL (Post-Boost [M24]) | 69 | 10
  Anti-PSC ≥ 2 µg/mL (Post-Boost [M24]): number analyzed (Participants) | 193 | 56
  Anti-PSC ≥ 2 µg/mL (Post-Boost [M24]) | 5 | 0
  Anti-PSC ≥ 0.3 µg/mL (Post-Boost [M48]): number analyzed (Participants) | 192 | 56
  Anti-PSC ≥ 0.3 µg/mL (Post-Boost [M48]) | 38 | 4
  Anti-PSC ≥ 2 µg/mL (Post-Boost [M48]): number analyzed (Participants) | 192 | 56
  Anti-PSC ≥ 2 µg/mL (Post-Boost [M48]) | 6 | 0

28. Primary Outcome: Concentration of Anti-PSC Antibodies
Description: as for outcome 22
Time Frame: At Year 4
Population: as for outcome 10
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | Menitorix Group | Meningitec Group
Number analyzed (Participants) | 197 | 58
µg/mL
  Anti-PSC (Pre-Primary): number analyzed (Participants) | 197 | 56
  Anti-PSC (Pre-Primary) | 0.19 [0.17 to 0.21] | 0.16 [0.15 to 0.18]
  Anti-PSC (Post-Primary): number analyzed (Participants) | 194 | 54
  Anti-PSC (Post-Primary) | 9.41 [8.55 to 10.36] | 11.88 [9.75 to 14.46]
  Anti-PSC (Pre-Boost): number analyzed (Participants) | 194 | 57
  Anti-PSC (Pre-Boost) | 0.76 [0.66 to 0.87] | 0.85 [0.66 to 1.09]
  Anti-PSC (Post-Boost [M1]) | 7.46 [6.55 to 8.49] | 3.76 [2.94 to 4.80]
  Anti-PSC (Post-Boost [M12]): number analyzed (Participants) | 161 | 45
  Anti-PSC (Post-Boost [M12]) | 0.48 [0.41 to 0.57] | 0.34 [0.26 to 0.45]
  Anti-PSC (Post-Boost [M24]): number analyzed (Participants) | 193 | 56
  Anti-PSC (Post-Boost [M24]) | 0.27 [0.23 to 0.30] | 0.19 [0.16 to 0.22]
  Anti-PSC (Post-Boost [M48]): number analyzed (Participants) | 192 | 56
  Anti-PSC (Post-Boost [M48]) | 0.21 [0.19 to 0.23] | 0.17 [0.15 to 0.19]

29. Primary Outcome: Number of Subjects With Anti-pertussis Toxoid (Anti-PT), Anti-filamentous Haemagglutinin (Anti-FHA) and Anti-pertactin (Anti-PRN) Antibody Concentrations Equal to or Above 5.0 ELISA Units Per Milliliter (EL.U/mL)
Description: The anti-pertussis toxoid, anti-filamentous haemagglutin, anti-pertactin activity was determined using an Enzyme-linked Immunosorbent Assay (ELISA).
Time Frame: At Year 2
Population: The ATP cohort for persistence Year 2 included all evaluable subjects who received 3 doses of vaccines in study NCT00258700, with available results for at least one tested antigen at Year 2. Persistence of anti-PT, anti-FHA and anti-PRN antibodies were evaluated for the UK subjects of Menitorix group and Meningitec group only
Measure: Number; unit: Subjects
Arm/Group | Menitorix Group | Meningitec Group
Number analyzed (Participants) | 67 | 23
Subjects
  Anti-PT Pre-Primary: number analyzed (Participants) | 64 | 18
  Anti-PT Pre-Primary | 11 | 3
  Anti-PT Post-Primary (M3): number analyzed (Participants) | 63 | 20
  Anti-PT Post-Primary (M3) | 63 | 20
  Anti-PT Post-Primary (M10): number analyzed (Participants) | 66 | 21
  Anti-PT Post-Primary (M10) | 34 | 10
  Anti-PT Pre-Boost | 8 | 3
  Anti-FHA Pre-Primary: number analyzed (Participants) | 65 | 19
  Anti-FHA Pre-Primary | 40 | 12
  Anti-FHA Post-Primary (M3): number analyzed (Participants) | 63 | 20
  Anti-FHA Post-Primary (M3) | 63 | 20
  Anti-FHA Post-Primary (M10): number analyzed (Participants) | 65 | 21
  Anti-FHA Post-Primary (M10) | 65 | 21
  Anti-FHA Pre-Boost: number analyzed (Participants) | 64 | 22
  Anti-FHA Pre-Boost | 47 | 13
  Anti-PRN Pre-Primary: number analyzed (Participants) | 64 | 19
  Anti-PRN Pre-Primary | 22 | 4
  Anti-PRN Post-Primary (M3): number analyzed (Participants) | 63 | 20
  Anti-PRN Post-Primary (M3) | 63 | 20
  Anti-PRN Post-Primary (M10): number analyzed (Participants) | 66 | 21
  Anti-PRN Post-Primary (M10) | 53 | 14
  Anti-PRN Pre-Boost | 34 | 7

30. Primary Outcome: Concentration of Anti-PT, Anti-FHA and Anti-PRN Antibodies
Description: Antibody concentrations for anti-pertussis toxoid, anti-filamentous haemagglutin and anti-pertactin C were expressed as geometric mean concentrations (GMC) with 95% confidence intervals (CI), given in EL.U/mL.
Time Frame: At Year 2
Population: as for outcome 29
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | Menitorix Group | Meningitec Group
Number analyzed (Participants) | 67 | 23
EL.U/mL
  Anti-PT Pre-Primary: number analyzed (Participants) | 64 | 18
  Anti-PT Pre-Primary | 3.2 [2.8 to 3.7] | 3.3 [2.4 to 4.6]
  Anti-PT Post-Primary (M3): number analyzed (Participants) | 63 | 20
  Anti-PT Post-Primary (M3) | 44.8 [39.1 to 51.2] | 40.1 [31.7 to 50.8]
  Anti-PT Post-Primary (M10): number analyzed (Participants) | 66 | 21
  Anti-PT Post-Primary (M10) | 4.9 [4.1 to 5.9] | 4.5 [3.3 to 6.1]
  Anti-PT Pre-Boost | 2.9 [2.6 to 3.2] | 3.0 [2.4 to 3.6]
  Anti-FHA Pre-Primary: number analyzed (Participants) | 65 | 19
  Anti-FHA Pre-Primary | 6.5 [5.2 to 8.2] | 7.8 [4.7 to 13.0]
  Anti-FHA Post-Primary (M3): number analyzed (Participants) | 63 | 20
  Anti-FHA Post-Primary (M3) | 223.5 [194.6 to 256.7] | 160.2 [123.1 to 208.6]
  Anti-FHA Post-Primary (M10): number analyzed (Participants) | 65 | 21
  Anti-FHA Post-Primary (M10) | 30.4 [25.7 to 35.9] | 25.8 [19.0 to 34.9]
  Anti-FHA Pre-Boost: number analyzed (Participants) | 64 | 22
  Anti-FHA Pre-Boost | 15.1 [9.5 to 24.0] | 20.3 [8.0 to 51.8]
  Anti-PRN Pre-Primary: number analyzed (Participants) | 64 | 19
  Anti-PRN Pre-Primary | 4.2 [3.4 to 5.2] | 3.1 [2.5 to 3.9]
  Anti-PRN Post-Primary (M3): number analyzed (Participants) | 63 | 20
  Anti-PRN Post-Primary (M3) | 116.3 [93.7 to 144.5] | 46.1 [31.0 to 68.5]
  Anti-PRN Post-Primary (M10): number analyzed (Participants) | 66 | 21
  Anti-PRN Post-Primary (M10) | 12.5 [9.5 to 16.2] | 6.6 [4.4 to 9.9]
  Anti-PRN Pre-Boost | 5.9 [4.5 to 7.7] | 4.3 [2.8 to 6.5]

31. Primary Outcome: Number of Subjects With Anti-PT, Anti-FHA and Anti-PRN Antibody Concentrations ≥ 5.0 EL.U/mL
Description: as for outcome 29
Time Frame: At Year 4
Population: as for outcome 10
Measure: Number; unit: Subjects
Arm/Group | Menitorix Group | Meningitec Group
Number analyzed (Participants) | 44 | 14
Subjects
  Anti-PT Pre-Primary: number analyzed (Participants) | 41 | 12
  Anti-PT Pre-Primary | 9 | 2
  Anti-PT Post-Primary (M3): number analyzed (Participants) | 42 | 11
  Anti-PT Post-Primary (M3) | 42 | 11
  Anti-PT Post-Primary (M10): number analyzed (Participants) | 44 | 13
  Anti-PT Post-Primary (M10) | 24 | 5
  Anti-PT Pre-Boost ( M32): number analyzed (Participants) | 43 | 14
  Anti-PT Pre-Boost ( M32) | 6 | 2
  Anti-PT Post-Boost ( M24): number analyzed (Participants) | 44 | 13
  Anti-PT Post-Boost ( M24) | 30 | 9
  Anti-FHA Pre-Primary: number analyzed (Participants) | 42 | 12
  Anti-FHA Pre-Primary | 27 | 9
  Anti-FHA Post-Primary (M3): number analyzed (Participants) | 42 | 11
  Anti-FHA Post-Primary (M3) | 42 | 11
  Anti-FHA Post-Primary (M10): number analyzed (Participants) | 44 | 13
  Anti-FHA Post-Primary (M10) | 43 | 13
  Anti-FHA Pre-Boost ( M32): number analyzed (Participants) | 41 | 13
  Anti-FHA Pre-Boost ( M32) | 29 | 10
  Anti-FHA Post-Boost ( M24): number analyzed (Participants) | 41 | 14
  Anti-FHA Post-Boost ( M24) | 41 | 14
  Anti-PRN Pre-Primary: number analyzed (Participants) | 41 | 12
  Anti-PRN Pre-Primary | 13 | 3
  Anti-PRN Post-Primary (M3): number analyzed (Participants) | 42 | 11
  Anti-PRN Post-Primary (M3) | 42 | 11
  Anti-PRN Post-Primary (M10): number analyzed (Participants) | 44 | 13
  Anti-PRN Post-Primary (M10) | 36 | 8
  Anti-PRN Pre-Boost ( M32): number analyzed (Participants) | 43 | 14
  Anti-PRN Pre-Boost ( M32) | 25 | 4
  Anti-PRN Post-Boost ( M24) | 43 | 14

32. Primary Outcome: Concentration of Anti-PT, Anti-FHA and Anti-PRN Antibodies
Description: Antibody concentrations for anti-pertussis toxoid, anti-filamentous haemagglutin and anti-pertactin were expressed as geometric mean concentrations (GMC) with 95% confidence intervals (CI), given in EL.U/mL.
Time Frame: At Year 4
Population: as for outcome 10
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | Menitorix Group | Meningitec Group
Number analyzed (Participants) | 44 | 14
EL.U/mL
  Anti-PT Pre-Primary: number analyzed (Participants) | 41 | 12
  Anti-PT Pre-Primary | 3.4 [2.8 to 4.1] | 3.4 [2.1 to 5.5]
  Anti-PT Post-Primary (M3): number analyzed (Participants) | 42 | 11
  Anti-PT Post-Primary (M3) | 45.2 [37.2 to 54.8] | 36.5 [26.1 to 51.1]
  Anti-PT Post-Primary (M10): number analyzed (Participants) | 44 | 13
  Anti-PT Post-Primary (M10) | 5.1 [4.1 to 6.4] | 3.9 [2.7 to 5.6]
  Anti-PT Pre-Boost ( M32): number analyzed (Participants) | 43 | 14
  Anti-PT Pre-Boost ( M32) | 3.0 [2.5 to 3.5] | 3.1 [2.3 to 4.1]
  Anti-PT Post-Boost ( M24): number analyzed (Participants) | 44 | 13
  Anti-PT Post-Boost ( M24) | 8.2 [6.1 to 10.9] | 7.2 [3.9 to 13.4]
  Anti-FHA Pre-Primary: number analyzed (Participants) | 42 | 12
  Anti-FHA Pre-Primary | 7.2 [5.2 to 10.0] | 9.1 [4.7 to 17.6]
  Anti-FHA Post-Primary (M3): number analyzed (Participants) | 42 | 11
  Anti-FHA Post-Primary (M3) | 229.9 [188.5 to 280.4] | 169.8 [127.0 to 227.0]
  Anti-FHA Post-Primary (M10): number analyzed (Participants) | 44 | 13
  Anti-FHA Post-Primary (M10) | 27.2 [22.1 to 33.5] | 22.8 [15.6 to 33.3]
  Anti-FHA Pre-Boost ( M32): number analyzed (Participants) | 41 | 13
  Anti-FHA Pre-Boost ( M32) | 16.7 [9.0 to 30.9] | 33.1 [9.6 to 113.8]
  Anti-FHA Post-Boost ( M24): number analyzed (Participants) | 41 | 14
  Anti-FHA Post-Boost ( M24) | 164.7 [119.4 to 227.1] | 66.8 [43.8 to 101.7]
  Anti-PRN Pre-Primary: number analyzed (Participants) | 41 | 12
  Anti-PRN Pre-Primary | 3.9 [3.1 to 4.9] | 3.1 [2.4 to 4.1]
  Anti-PRN Post-Primary (M3): number analyzed (Participants) | 42 | 11
  Anti-PRN Post-Primary (M3) | 135.6 [106.0 to 173.4] | 50.4 [26.0 to 97.6]
  Anti-PRN Post-Primary (M10): number analyzed (Participants) | 44 | 13
  Anti-PRN Post-Primary (M10) | 12.2 [8.9 to 16.7] | 5.6 [3.6 to 8.8]
  Anti-PRN Pre-Boost ( M32): number analyzed (Participants) | 43 | 14
  Anti-PRN Pre-Boost ( M32) | 6.6 [4.5 to 9.5] | 4.9 [2.4 to 9.8]
  Anti-PRN Post-Boost ( M24) | 102.8 [67.1 to 157.3] | 23.4 [15.1 to 36.2]

33. Primary Outcome: Number of Subjects With Serious Adverse Events (SAEs)
Description: A SAE was defined as any medical occurrence that resulted in death, was life-threatening, required hospitalization or prolongation of hospitalization, resulted in disability/incapacity in a subject. AE(s) considered as SAE(s) also included invasive or malignant cancers, intensive treatment in an emergency room or at home for allergic bronchospasm, blood dyscrasias or convulsions that did not result in hospitalization, as per the medical or scientific judgement of the physician. Any = Occurrence of a SAE, regardless of relationship to vaccination.
Time Frame: Up to Month 12 (Booster vaccination)
Population: The Booster Total Vaccinated Cohort included all subjects who received the booster dose during study NCT00258700.
Measure: Number; unit: Subjects
Arm/Group | Menitorix Group | Meningitec Group
Number analyzed (Participants) | 359 | 117
Subjects | 0 | 0

34. Primary Outcome: Number of Subjects With SAE(s)
Description: as for outcome 33
Time Frame: Up to Month 24 (Booster vaccination)
Population: The Booster Total Vaccinated Cohort included all subjects who received the booster dose during study NCT00258700.
Measure: Number; unit: Subjects
Arm/Group | Menitorix Group | Meningitec Group
Number analyzed (Participants) | 359 | 117
Subjects | 0 | 0

35. Primary Outcome: Number of Subjects With SAE(s)
Description: as for outcome 33
Time Frame: Up to Month 48 (Booster vaccination)
Population: The Booster Total Vaccinated Cohort included all subjects who received the booster dose during study NCT00258700.
Measure: Number; unit: Subjects
Arm/Group | Menitorix Group | Meningitec Group
Number analyzed (Participants) | 359 | 117
Subjects | 1 | 0

36. Primary Outcome: Number of Subjects With SAE(s)
Description: as for outcome 33
Time Frame: Within (31-Days) at Year 2
Population: The Total Cohort Year 2 included all vaccinated subjects in the booster study NCT00258700, who came back for the Year 2 follow-up and also all subjects of Meningitec+Hiberix Group who were enrolled and vaccinated at Visit 2 in study NCT00454987 (i.e. 40-43 months of age).
Measure: Number; unit: Subjects
Arm/Group | Menitorix Group | Meningitec Group | Meningitec+Hiberix Group
Number analyzed (Participants) | 70 | 23 | 72
Subjects | 1 | 0 | 0

ADVERSE EVENTS:
Time Frame: SAEs: from booster study NCT00258700 until the end of the persistence study (M48).
Description: No information about unsolicited adverse events was collected during this study. SAEs were collected on the total number of subjects in the NCT00258700 study (476), which included the subjects enrolled in this NCT00454987 study.
Arm/Group | Menitorix Group | Meningitec Group | Meningitec+Hiberix Group
All-Cause Mortality (participants affected / at risk) | 0/359 | 0/117 | 0/74
Serious Adverse Events (participants affected / at risk) | 2/359 | 0/117 | 0/74
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Menitorix Group (N=359) | Meningitec Group (N=117) | Meningitec+Hiberix Group (N=74)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1/70 | 0/23 | NA
Pyrexia (General disorders) | 1 | 0 | NA

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.